CLINICAL TRIAL: NCT00744588
Title: Stress, HPA Dysfunction, and Relapse in Alcoholism
Brief Title: Stress, Hypothalamic-pituitary-adrenal (HPA) Dysfunction, and Relapse in Alcoholism
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Dallas VA Medical Center (U.S. Federal Agency); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Bryon H Adinoff, Professor, University of Texas Southwestern Medical Center
Other Study IDs: AA016668; U01AA016668 (NIH)
Record Dates: First submitted 2008-06-19; First posted 2008-09-01 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Alcohol Dependence
Keywords: substance abuse; alcohol dependence; hypothalamic-pituitary-adrenal (HPA) system; cosyntropin; corticotropin-releasing Hormone (CRH); pituitary-adrenal system; stress; trauma; neurosteroids; cortisol; relapse
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Phenylketonurias; Wounds and Injuries; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum plasma whole blood urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- alcohol dependence: Alcohol-dependent subjects currently being treated in an inpatient treatment facility.

SUMMARY:
This proposal is part of the INIA Stress Consortium. This study will

1. explore the contributions of lifetime trauma, recent stress, and alcohol use on stress-hormone axis disruption in treatment seeking, one-month abstinent, alcohol-dependent subjects
2. assess the combined contributions of stress-hormone axis disruption and episodic stress on the risk of prospective drinking following treatment
3. determine the role of neurosteroids in alcohol use.

DETAILED DESCRIPTION:
The hypothalamic-pituitary-adrenal (HPA) system is suggested as a key biologic link in stress-induced relapse. The HPA axis provides a regulatory feedback network between the brain and the body's behavioral and physiologic responses to stress, recovery, and adaptation. Both trauma and chronic alcohol use produce persistent disturbances in the HPA response to stress. The chronic use of alcohol may also impair the stress-induced release of neurosteroids, compounds that directly modulate central nervous system activity. Thus, altered cortisol and neurosteroid responsiveness during abstinence may impair the central nervous system's ability to mount an appropriate response to environmental stressors, heightening the probability of relapse. However, the relationship between stress, relapse, and HPA axis disturbances remains tentative. In the proposed study, the investigators will assess the contribution of trauma, stress, and alcohol use upon pituitary-adrenocortical functioning in alcohol dependence. The relative contribution of adrenocortical disruption and episodic stress to prospective drinking behaviors will then be determined.

Hypothesis: We hypothesize (1) that lifetime trauma, recent stress, and chronic alcohol use will additively contribute to HPA axis disruption, (2) alterations in glucocorticoid and neurosteroid release as well as episodic stress will predict a return to drinking.

Methods: One hundred treatment-seeking, one-month abstinent, alcohol-dependent subjects will be studied. Standardized assessments will be used to assess childhood and adult trauma as well as recent (six months) stress. Pituitary-adrenal (including ACTH (adrenocorticotropin), cortisol, and neurosteroids) responses to both neuroendocrine [ovine corticotropin releasing hormone (oCRH), cosyntropin, and dexamethasone] and experiential (public speaking) challenges will be measured. Drinking behavior and episodic stress will be prospectively assessed for six months following neuroendocrine assessment.

Significance: If our hypotheses are supported, a definitive connection between previous trauma, biological stress response mechanisms, and ongoing stress upon prospective drinking behavior will be demonstrated. The identification of a specific biologic mechanism that underlies this association will provide a fertile framework for the development of targeted pharmacological interventions to decrease relapse in this vulnerable population. In addition, elucidating the concurrent contributions of stress-response biologic systems and externals stressors will provide the therapist and patient with a constellation of specific risk factors for focused treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of alcohol dependence

Exclusion Criteria:

* Medical or psychiatric disorders that may effect stress-hormone axis functioning.
* Medications that may effect stress-hormone axis functioning.
* English speaking.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Inpatient treatment facility for substance use disorders.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2007-08; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Examine the contributions of previous trauma, recent stress, and chronic alcohol use to the stress-hormone axis reactivity in one-month abstinent alcohol-dependent subjects. | one month

SECONDARY OUTCOMES:
Assess the ability of stress-hormone axis reactivity and ongoing stress to predict subsequent drinking behavior following treatment discharge. | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Bryon Adinoff, MD, Principal Investigator — UT Southwestern Medical Center at Dallas and VA North Texas Health Care System
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States